CLINICAL TRIAL: NCT03351582
Title: Family Support for Grief and Communication
Brief Title: Grief and Communication Family Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ersta Sköndal University College (Other)
Responsible Party: Principal Investigator, Josefin Sveen, Associate professor in medical psychology, Ersta Sköndal University College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DRN 2016/1192/31/1
Record Dates: First submitted 2017-11-14; First posted 2017-11-24 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Grief; Communication
Keywords: family therapy; psychological health
MeSH Terms: conditions — Communication; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Grief and Communication One Session (Experimental): Group one will meet with a family therapist for one 90 minute session where the main focus will be on providing psychoeducation on grief and communication to both children and parents. This arm receives only the first session of the grief and communication family intervention.
  Interventions: Behavioral: Grief and Communication Family Intervention
- Grief and Communication Three Sessions (Experimental): Thie Group will receive all three sessions of the grief and communication family intervention.
  Interventions: Behavioral: Grief and Communication Family Intervention
- Control (No Intervention): Group three will be the control group and will not receive the grief and communication family intervention.

INTERVENTIONS:
Behavioral: Grief and Communication Family Intervention — This intervention is an integrative approach which uses techniques from systemic family therapy as well as cognitive behavioral therapy.
  Arms: Grief and Communication One Session; Grief and Communication Three Sessions

SUMMARY:
The overall purpose of this project is to evaluate the effects of a family therapy intervention for grieving families with children. The main outcome variable is family communication.

DETAILED DESCRIPTION:
The intervention study will test a supportive family therapy intervention for families where a parent has died from cancer between 2013 and 2015. This will be a randomized controlled trial where participants are assigned to one of three groups using a random number sequence generated by a computer program with approximately 25 families in each intervention group.

Group one will meet with a family therapist for one 90 minute session where the main focus will be on providing information through psychoeducation on grief and communication to participants.

Group two will participate in a family therapy intervention comprised of three 90 minute sessions. participants will receive the same psychoeducation as group one and will also work with the family therapist to enhance family communication and process their grief. The 3 sessions are manual based.

Group three will be the control group and will not meet with a family therapist.

Participants will be asked if their sessions with the family therapist can be tape-recorded, but do not have to consent to this in order to participate. Approximately 6 participants need to be recorded in order to ensure that the family therapists are covering the same topics and giving the same information to all participants. In this way we can ensure that the method of intervention is the same no matter which therapist is delivering the intervention thereby validating the method of intervention.

Follow up will occur 1 month and 6 months after the intervention has ended. Each participant will fill in a short questionnaire regarding grief and Communication. Validated instruments will also be included in the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Participants are families with Children ages 3-19 who have completed our questionnaire study and have responses indicating that one or more family members have symptoms of complicated grief or a negative pattern of communication within the family. All family members who live in the same home may participate in the family therapy intervention including new partners or step children. It is up to the family to decide which family members will be included.

Exclusion Criteria:

* Participants must reside in Stockholm, Sweden during data collection, speak and understand written and spoken Swedish.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Parent-Adolescent Communication Scale | Change from baseline score at one month, six month, and 18 month follow up
  questionnaire- scores between 20-100 with higher scores indicating better family communication.

SECONDARY OUTCOMES:
The Prolonged Grief Disorder Inventory PG-13 | Change from baseline score at one month, six month, and 18 month follow up
  questionnaire- scores range between 11-55 higher scores indicate more symptoms of prolonged grief
Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Change from baseline score at one month, six month, and 18 month follow up
  questionnaire-The items are rated on a 5-point scale with response descriptors 0 ''not at all'' to 4 ''extremely''. Total scores range from 0 to 80 and a preliminary cut-off score of 33 is suggested as indicating PTSD
Montgomery-Åsberg Depression Rating Scale | Change from baseline score at one month, six month, and 18 month follow up
  questionnaire-The MADRS was used to assess symptoms of depression. It consists of 9 items. Each item is scored on a 6-point Likert scale. The total score is calculated by summing the answers of the nine items, ranging between 0 and 54 and a higher score indicates a greater risk of depression. Cut off is usually put at 10 for mild depression, 20 for moderate depression and >34 for severe depression
The Generalized Anxiety Disorder scale (GAD-7) | Change from baseline score at one month, six month, and 18 month follow up
  The GAD-7 was used to assess symptoms of anxiety. It consists of 7 items, scored on a 4-point scale to the response categories from "not at all" to "nearly every day", and adding together the scores for the seven questions. Total scores of 5, 10, and 15 are taken as the cut-off for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or more
The Strengths and Difficulties Questionnaire (SDQ) | Change from baseline score at one month, six month, and 18 month follow up
  questionnaire- subscale externalizing symptoms scores range from 0-20 with higher scores indicating more internalizing problems. Externalizing subscale scores range from 0-20 with higher scores indicating more externalizing problems.
Trauma cognitions checklist | Change from baseline score at one month, six month, and 18 month follow up
  Parent report of children's PTSD symptoms. Scores range from 9-27 with higher scores indicating more PTSD symptoms
Rosenberg self-esteem scale | Change from baseline score at one month, six month, and 18 month follow up
  questionnaire- scores range between 10-40 with higher scores indicating higher self-esteem

CONTACTS AND LOCATIONS:
Overall Officials: Josefin Sveen, PhD, Principal Investigator — Ersta Sköndal University College
Locations (1):
- Private clinic, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No